CLINICAL TRIAL: NCT07375485
Title: Multifaceted Implementation Program for Occupational Therapy Practitioners Addressing Anxiety and Depressive Symptoms in Home and Community Care
Brief Title: Occupational Therapy for Mental Health and Engagement in Neurorehabilitation
Acronym: OT for ME
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Rehab Without Walls Neurorehabilitation (Unknown); American Occupational Therapy Foundation (Other)
Responsible Party: Principal Investigator, Janell Pisegna, Assistant Professor, Colorado State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #: 6989
Record Dates: First submitted 2026-01-03; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Acquired Brain Injury; Mental Health; Depressive Symptoms; Anxiety Symptoms; Loneliness
Keywords: Occupational therapy; Mental health; Acquired brain injury; Implementation
MeSH Terms: conditions — Brain Injuries; Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occupational therapy practitioners (Experimental): OTPs will complete training and coaching sessions on evidence-based OT mental health screening (anxiety and depressive symptoms and loneliness) and intervention practices (cognitive behavioral therapy, problem-solving therapy, motivational interviewing, behavior change, and self-regulation), receive job and decision aid templates, attend monthly check-insas a team and with clinical experts in OT mental healthcare, and fidelity monitoring and observation. Additional strategies may be identified through interviews or focus groups by tailoring implementation strategies further to the local context. Interdisciplinary team members will only undergo the training and share their experiences and perceptions of OT's role in mental health during neurorehabilitation.
  Interventions: Behavioral: Multifaceted implementation program

INTERVENTIONS:
Behavioral: Multifaceted implementation program — OTPs will complete training and coaching sessions on evidence-based OT mental health screening (anxiety and depressive symptoms and loneliness) and intervention practices (cognitive behavioral therapy, problem-solving therapy, motivational interviewing, behavior change, and self-regulation), receive job and decision aid templates, attend monthly check-insas a team and with clinical experts in OT mental healthcare, and fidelity monitoring and observation. Additional strategies may be identified by the OT practitioners in the study through interviews or focus groups, allowing for further tailoring of implementation strategies to the local context.

SUMMARY:
Changes in mental health are common after acquired brain injury (ABI), defined as any traumatic or non-traumatic injury to the brain after birth, affecting approximately 1 in 3 adults with ABI. Occupational therapy (OT) practitioners are uniquely qualified to contribute to addressing how mental and physical health influence engagement in activities of daily living, yet many OT practitioners working in neurorehabilitation do not implement recommended evidence-based mental health screening or intervention. This study aims to test a comprehensive implementation program for integrating evidence-based mental healthcare into OT rehabilitation services for people with ABI. The study will be conducted with OT practitioners working in home and community neurorehabilitation settings. The focus of the study is to better understand strategies to help OT practitioners adopt and implement evidence-based mental healthcare into routine practice. By doing so, the study aims to improve neurorehabilitation care delivery and promote positive mental health and community engagement among people with ABI.

DETAILED DESCRIPTION:
This Hybrid Type 3 convergent mixed methods pilot study examines implementation processes, practitioner experiences, and stakeholder perspectives associated with participation in a multifaceted implementation program designed to support OTPs in addressing mental health among adults with ABI in home and community-based care.

Participating OTPs complete a virtual, self-paced, five-module educational training focused on evidence-based mental health screening and intervention strategies relevant to ABI. Additional implementation support activities include periodic check-ins, mentoring and coaching as part of routine clinical practice, fidelity monitoring, and audit and feedback through electronic health record review.

Aim 1. Describe reach, adoption, implementation experiences, and maintenance of mental health-related occupational therapy practices among OTPs participating in a multifaceted implementation training in home and community-based neurorehabilitation.

Aim 2. Explore implementation mechanisms and contextual factors influencing observed implementation experiences, informed by the Practical, Robust Implementation and Sustainability Model (PRISM).

Aim 3. Describe perspectives of key stakeholders, including interdisciplinary team members, administrators, and people with ABI, regarding their experiences of OT addressing mental health.

The primary outcomes of the study are changes in OT practitioners' knowledge, self-efficacy, and mental health practice skills (defined according to the Reach Effectiveness Adoption Implementation and Maintenance [RE-AIM] Model). These outcomes will be assessed through electronic health record review, fidelity monitoring, surveys, and focus groups.

Interdisciplinary stakeholders, including social work, neuropsychology, administrative leadership, patients with ABI and caregivers will participate in focus groups and interviews to provide perspectives on feasibility, acceptability, and perceived impact of the training within the clinical setting.

ELIGIBILITY:
Inclusion criteria are at the level of the therapist:

* State-licensed occupational therapists (OTs) or occupational therapy assistants (OTAs) in the United States
* OTs or OTAs who work in home or community neurorehabilitation practice settings and treat adults (18 years of age or older) with acquired brain injury (defined as any traumatic or non-traumatic injury to the brain after birth)

Exclusion Criteria:

* OTs or OTAs without a state license to practice OT
* OTs or OTAs who do not work in home or community neurorehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Implementation outcomes | 24 months
  The primary outcome of this study is the adoption of evidence-based mental health screening and intervention practices among occupational therapy practitioners after participating in a multifaceted implementation program.
  We have defined adoption as a dichotomous outcome (adopted vs. did not adopt), with the a priori established benchmark for adoption as the observed use of evidence-based mental health screening tools and intervention practices with 90% of clients in 10 or more sessions across the client's length of stay.
  We will measure adoption using directed content analysis of electronic health record data, on-site observations, and self-reported use of screening and intervention practices from qualitative focus groups and interviews.

SECONDARY OUTCOMES:
Identify implementation mechanisms and factors influencing implementation outcomes | 24 months
  The secondary outcome of this study is to understand factors that influenced the adoption of evidence-based mental health screening and intervention practices among occupational therapy practitioners after participation in a multifaceted implementation program.
  Factors influencing the adoption of mental health screening and intervention practices will be measured qualitatively through the identification of themes that influence whether practitioners adopt the mental health screening tools and interventions. We will thematically analyze focus group and interview transcripts with inductive and deductive (from the Practical, Robust Implementation and Sustainability Model [PRISM] and use of a codebook) codes to identify the themes.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rehab Without Walls Denver, CO, Denver, Colorado
  - Colorado State University, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: No
A small number of sites pose risks to participant privacy and confidentiality, and risk for identification. IPD would only be shared with a data use agreement between all relevant parties.